CLINICAL TRIAL: NCT02438514
Title: Biological Biomarkers in MOMS Partnership
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1410014845
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Biological Sample Collection — Anthropomorphic biomarkers including height, weight, heart rate, and blood pressure will be taken for each participating mother and child by a research assistant trained to accurately perform these procedures.
  Blood spots will be collected in finger stick proficiency, using trigger activated lancets to administer finger sticks.
  Each participating mothers and child will provide a saliva sample using Oragene DNA saliva collection kits

SUMMARY:
The investigators propose to evaluate the potential utility of stress-related biomarkers obtained via dried blood spots (DBS) and retinal scans by collecting new data from mothers and children within the New Haven MOMS Partnership, a well-established community-partnered research setting. The proposed research could greatly advance the application of stress-related biomarkers within community-based research by increasing our understanding of how stress, trauma, and depression influence biology in childhood and adulthood, as measured using minimally-invasive approaches.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult mothers (age 21 or older) of at least one biological child mothers must be able to answer three verification questions to confirm they are the biological parent of their child

Exclusion Criteria:

* Non-english speakers
* Women not able to provide informed consent and with no biological children
* Mothers under the age of 21

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low-income, racially and ethnically diverse, un- or under-employed, biological mothers of children in New Haven.
  Primary source of recruitment will be the screening/needs assessment from our affiliated MOMS Partnership protocol, however, we will actively respond to inquiries from any preliminarily eligible biological mother in the New Haven community who expresses interest in the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2019-01 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Number of Mother-Child Dyads Who Complete Assessments & Biological Samples | End of study (approximately 5 years)
  Feasibility outcome
Telomere Length | At baseline-After 90 minutes
  Telomere length will be measured using an adapted method of the Cawthon Telomere Assay
Advanced Glycation End Products (AGEs) | At baseline-After 90 minutes
  AGEs or (advanced glycation endproducts) will be measured using a painless non- invasive retinal scanning device that measures autofluorescence of the crystalline lens of the eye

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States